CLINICAL TRIAL: NCT06817200
Title: The Effect of Amantadine as add-on Therapy for Motor Fluctuations in Advanced Parkinson's Disease: a Randomized Double-blinded Placebo-controlled Trial
Acronym: AMANT-OFF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/23/0372; 2023-509728-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson's disease; clinical trial; Motor fluctuations; Amantadine
MeSH Terms: conditions — Parkinson Disease | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amantadine (Experimental): Amantadine will be administered at the dose of 100 mg t.i.d or b.i.d. (if t.i.d. is not tolerated) over 12 weeks, after a period of 3 weeks of titration.
  The study treatment will be stopped after a dose decrease of 100 mg / day every 3 days.
  Interventions: Drug: Amantadine (100mg) as add on therapy.
- Placebo (Placebo Comparator): Placebo tablets will be also administered b.i.d. or t.i.d over 12 weeks after a period of 3 weeks of titration. Placebo tablets will be indistinguishable from amantadine ones.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine (100mg) as add on therapy. — Amantadine will be administered at the dose of 100 mg t.i.d or b.i.d. (if t.i.d. is not tolerated) over 12 weeks, after a period of 3 weeks of titration.T he study treatment will be stopped after a dose decrease of 100 mg / day every 3 days.
  Arms: Amantadine
Drug: Placebo — Placebo tablets will be also administered b.i.d. or t.i.d over 12 weeks after a period of 3 weeks of titration. Placebo tablets will be indistinguishable from amantadine ones.
  Arms: Placebo

SUMMARY:
Motor fluctuations are identified as the most challenging symptoms by parkinson disease patients. A recent post-hoc analysis of ADS-5012 trials (new formulation of ER Amantadine), revealed a significant improvement in OFF-time. No randomized clinical trial has ever specifically investigated to date the effect of amantadine IR on motor fluctuations. The main objective of this study is to evaluate the effect of amantadine (300 mg/day) as add-on therapy for the treatment of motor fluctuations (Off-time) in advanced Parkinson's disease patients versus placebo after 3 months of treatment.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common age-related neurodegenerative disorder. Up to 50% of parkinson disease patients develop mild motor fluctuations (OFF-time) within 2 years of initiating levodopa therapy, increasing up to 70% of patients after 9 years. Motor fluctuations are identified as the most challenging symptoms by parkinson disease patients and considered as a key clinical unmet need for advanced parkinson disease patients. Amantadine has been approved by the FDA in 1973 for the "treatment of parkinson disease". It has a unique pharmacodynamic profile with both a dopaminergic and an anti-glutamatergic effect, which are related to its anti-parkinsonian and anti-dyskinetic action. In 2017, the FDA approved 2 new Amantadine extended release (ER) formulations for dyskinesia treatment, ADS-5012 and OS-320. In 2021 post-hoc analysis of ADS-5012 trials, revealed a significant improvement in OFF-time (1 h of reduction vs. placebo). These findings led to the FDA granting amantadine ER an additional indication as add-on treatment to levodopa for the management of motor fluctuations. No randomized clinical trial has ever specifically investigated to date the effect of amantadine Immediate Release on motor fluctuations. We hypothesize that the double action of amantadine could allow this drug to be effective in the treatment of motor fluctuations, without increasing dyskinesia. Parkinson disease patient with motor fluctuations will be included and followed up in this study. After 3 to 4 weeks of titration, patients will receive stable dose of amantadine (up to 300 mg/day) or matching placebo during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease diagnosis in agreement with the MDS criteria (Postuma et al., 2015) for at least 3 years HY 2-3 in Med ON condition Age: 30-80 years Signs of motor fluctuations for at least 4 weeks before screening, with a mean total awake time in the off state of at least 2 h, including morning akinesia despite anti-parkinsonian drug adjustment (best medical treatment)" Amantadine naïve (all other oral add-on treatments for motor fluctuations are allowed) Concomitant anti-Parkinson drug use should be stable for at least 4 weeks prior to screening Patients affiliated or beneficiary of a social security scheme. Patients who signed the written informed consent form. Patients in capacity to complete Hauser diaries

Exclusion Criteria:

Severe or unpredictable periods in the Off-state, or both; Clinically significant and unstable cardiovascular disease, psychiatric illness (including major depression, dementia, impulse control, disorders, and suicide ideation), or any other medical disorder that might have placed the patient at increased risk; Patient with behavioral disorder, ECMP item ≥ 3 Patients previously submitted to advanced treatments: subcutaneous continuous apomorphine infusion, deep brain stimulation and levodopa-carbidopa intestinal gel; Patients with cognitive impairment (Mini Mental Status Examination < 26) Patients with a diagnosis of atypical parkinsonism (Progressive supranuclear Palsy, Multiple system atrophy, Lewy Body Dementia or Cortico-basal degeneration) Patients having any contraindication to amantadine treatment (see Summary of Product characteristic in the Appendix: known hypersensitivity to drugs of the amantadine class or any of the components, combination with anti-emetic neuroleptics, patient with a history of epilepsy, confusional state, hallucinations or severe psychoneurotic state not controlled by treatment, patient with a history of congestive heart failure or peripheral oedema, patient with a history of skin eczema) A history of neuroleptic malignant syndrome or nontraumatic Rhabdomyolysis; renal failure and renal insufficiency (creatinine > 150 µmol/L) states of agitation or confusion delirious syndromes or exogenous psychosis in the anamnesis Has received any other investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening or plans to use an investigational drug (other than the study intervention) during the study Pregnant female subjects or potential childbearing female participant without highly effective contraception

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
the change in motor fluctuation (Off-time) | 3 months
  The primary outcome of this study is the change from baseline to end-point (3 months) in motor fluctuation (Off-time) as assessed by the Hauser diaries (average of 3 consecutive days).

SECONDARY OUTCOMES:
The rate of Off-time responders | 3 months
  The change from baseline to end-point (3 months) of the rate of Off-time responders
The change of the mean score of MDS-UPDRS part IV | 3 months
  The change from baseline to end-point (3 months) of The mean score of Movement disorders society - Unified Parkinson's disease rating scale (MDS-UPDRS part IV)
The change of the mean score of UDysRS part 2A | 3 months
  The change from baseline to end-point (3 months) of the mean score of UDysRS part 2A
The change of the mean score of New freezing of gait questionnaire | 3 months
  The change from baseline to end-point (3 months) of the mean score of New freezing of gait questionnaire
The change of the mean score of Fatigue Severity Scale | 3 months
  The change from baseline to end-point (3 months) of the mean score of Fatigue Severity Scale
The change of the mean score of MDS-UPDRS Part I-II-III | 3 months
  The change from baseline to end-point (3 months) of the mean score of Movement disorders society - Unified Parkinson's disease rating scale (MDS-UPDRS Part I-II-III)
The change of the mean score of PDQ-39 | 3 months
  The change from baseline to end-point (3 months) of the mean score of Parkinson's Disease Questionnaire (PDQ-39)
The safety of amantadine | 3 months
  The safety of amantadine, expressed as: the percentage of Adverse Events, of severe Adverse Events, of serious Adverse Events and of patients' discontinuation due to Adverse Events, all over the three months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Toulouse, Toulouse, France